CLINICAL TRIAL: NCT05830565
Title: Survey on the Management of Occasional or Anticipatory Stress by Consumers of a Food Supplement Based on L-theanine, Passionflower and Rhodiola Extracts and Satisfaction With This Supplementation
Brief Title: Management of Occasional or Anticipatory Stress by Consumers of a Food Supplement
Acronym: MELIM
Status: Completed | Type: Observational
Sponsor: Larena SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: PIL-RIPH3-MELIM-023
Record Dates: First submitted 2023-03-07; First posted 2023-04-26 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-05

CONDITIONS: Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Food Supplement: Single dose of food Supplement Based on L-theanine, Passionflower and Rhodiola Extracts

SUMMARY:
Volunteers will fill out an initial questionnaire which will describe their current situation, their pathologies and current treatments, their medical history.

Finally, they will complete three questionnaires on the day of their stressful event which will describe their state of stress just before taking the product, 20 minutes after taking the product; their tolerance and satisfaction with the product will be described at the end of the day.

DETAILED DESCRIPTION:
Participants in the survey will come from a panel of volunteers. They will be contacted via an email proposing the survey accompanied by a selection questionnaire. Eligible volunteers will be called by the clinical investigation center to confirm their participation.

Volunteers will fill out an initial questionnaire which will describe their current situation (sex, age, family and professional situation, cigarette consumption), their pathologies and current treatments, their medical history (disorders related to sleep, stress, anxiety, burnout, depression or other mental disorders).

Finally, they will complete three questionnaires on the day of their stressful event which will describe their state of stress just before taking the product, 20 minutes after taking the product; their tolerance and satisfaction with the product will be described at the end of the day.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* PSS Questionnaire (Perceived Stress Scale) ≥ 14
* Believing that they could be exposed to a stressful event in the next 2 months

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Currently taking a treatment from the following list: antihypertensives, immunosuppressants, antidepressants/barbiturates, anxiolytics, vitamin K antagonists (warfarin, acenocoumarol, fluindione), miconazole, anticonvulsants (carbamazepine, phenobarbital, phenytoin, oxcarbazepine...) and/or anti -infectious (rifampicin, rifabutin, efavirenz, nevirapine, griseofulvin)
* With diabetes, autoimmune disease or hypotension
* Currently taking a medication or dietary supplement that may affect mood, stress, sleep or anxiety
* Currently using products containing any of the following ingredients: hawthorn, ashwagandha (Withania somnifera), bacopa monnieri, black grass, holy basil (Ocimum sanctum), fig buds, CBD, Eleutherococcus, Eschscholtzia, ginseng, griffonia, hops, oil lavender essential oil, marjoram essential oil, lavender hydrolyzate, milk protein hydrolyzate (Lactium), inositol, magnesium, lemon balm, St. John's wort, angelica orange, passionflower, rhodiola, saffron, theanine, asparagus stalk, tryptophan, valerian
* Having known allergies to the ingredients of the product (theanine, rhodiola, passionflower and lavender)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult believing that they could be exposed to a stressful event in the next 2 months
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Evolution of level of felt stress before and after product intake | Before and 20 minutes after product intake
  Change in stress VAS (visual analogue scale), minimum = 0 and maximum = 10 higher score means a worse outcome

SECONDARY OUTCOMES:
Percentage of stress enhancement responders | Before and 20 minutes after product intake
  Percentage of volunteers with a decrease in the VAS scale
Evolution of level of felt stress | stress usually felt, just before product intake, 20 minutes after product intake and before midnight
  Change in stress VAS (visual analogue scale), minimum = 0 and maximum = 10 higher score means a worse outcome
Evolution of stress-related signs before and after product intake | Before and 20 minutes after product intake
  Percentage of volunteers with a decrease in the stress-related signs VAS scales
Percentage of stress-related signs enhancement responders | Before and 20 minutes after product intake
  Percentage of volunteers with a decrease in the stress-related signs VAS scales
EvaluatIon of the organoleptic properties | Before midnight
  Evaluation with a Likert scale, minimum = very unpleasant and maximum = pleasant higher score means a best outcome
satisfaction felt by volunteers | Before midnight
  Evaluation with a Likert scale, minimum = not effective and maximum = very effective higher score means a best outcome
Adverse events | Before midnight
  Number and type of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Carole Perrin, Principal Investigator — CEN
Locations (1):
- Cen Experimental, Dijon, France